CLINICAL TRIAL: NCT04665362
Title: A Single-arm Study to Evaluate the Safety and Efficacy of Recombinant Oncolytic Virus M1 (M1-c6v1) Combined With Anti-PD-1 Antibody SHR-1210 and Apatinib for Treatment of Patients With Advanced / Metastatic Hepatocellular Carcinoma
Brief Title: IIT Study of M1-c6v1 Combined With SHR-1210 and Apatinib in Patients With HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liang Peng (Other)
Collaborators: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Liang Peng, Principle Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-C02
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Advanced/Metastatic Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M1-c6v1 combined with SHR-1210 and Apatinib (Experimental): Single-arm
  Interventions: Drug: Recombinant oncolytic virus M1, anti PD-1 antibody, Apatinib

INTERVENTIONS:
Drug: Recombinant oncolytic virus M1, anti PD-1 antibody, Apatinib — Drug: Recombinant oncolytic virus M1
  Recombinant oncolytic virus M1 is administered intravenously 1×109 CCIC50 once daily on day1-5, every 28 day cyle.
  Other name：M1-c6v1
  Drug：Anti-PD-1 antibody
  Anti-PD-1 antibody is administered intravenously 200 mg once every 2 weeks.
  Other names：SHR-1210, Camrelizumab
  Drug: Apatinib
  Apatinib is administered orally 250mg once daily.
  Other name: Apatinib

SUMMARY:
This is a single arm and open-label phase I trial to evaluate the safety, tolerability and efficacy of the oncolytic virus M1 （M1-c6v1）(iv 1×109 CCIC50, 1 dose per day, on day 1-5 each 28 day cycle) combined with anti-PD-1 antibody SHR-1201 (iv, 200 mg, once every two weeks) and Apatinib (po. 250 mg qd ) in the patients with advanced/metastatic hepatocellular carcinoma. 10 participants will be sequentially enrolled. The treatment duration is 12 months. All patients continue combination treatment until disease progression, unacceptable toxicity, death, or discontinuation for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old, both genders.
2. To be confirmed to meet the clinical diagnosis standard, histologically or cytologically confirmed with hepatocellular carcinoma
3. Life expectancy of at least 3 months.
4. Patients was not received any systemic therapies to HCC.
5. For patients with advanced hepatocellular carcinoma, liver function status Child-Pugh Class A or B (score<=7).
6. HCC staging is evaluated according to Diagnostic and therapeutic criteria for liver cancer (2019 Edition, National health commission, P.R.A)

   * a: with vascular invasion and no extrahepatic metastasis, no matter the tumor condition; Child-Pugh A/B；PS 0~2.
   * b: with extrahepatic metastasis, no matter the tumor condition and vascular invasion; Child-Pugh A/B；PS 0~2, not eligible for surgical and/or locoregional therapies.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2.
8. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria (The long diameter of the lesion on spiral CT scan was more than or equal to 10 mm or the short diameter of enlarged lymph node was more than or equal to 15 mm).
9. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment)as determined by:

   ① Blood system: Hemoglobin ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L.

   ② Liver function: Serum total bilirubin (TBIL)≤2 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤5×upper limit of normal(ULN), Serum albumin ≥ 28 g/L; Alkaline phosphatase(ALP) ≤5×ULN;

   ③ Kidney function: Calculated creatinine clearance (CrCl) > 50 mL/min (Cockcroft-Gault formula will be used to calculate CrCl); Creatinine (Cr) ≤ 1.5×ULN; Urine protein <2+ or Baseline of urine protein ≥ 2+ and 24h urinary protein quantity ≤ 1g.

   ④ Coagulation function: International Normalized Ratio (INR) or Activated partial thromboplastin time (APTT) ≤ 1.5×ULN
10. Reproductive subjects (male and female) must agree to use effective birth control measures with their partners for at least 180 days after the last medication.
11. Volunteer to participate in clinical research; fully understand and be able to sign the informed consent form (ICF); willing to follow and have the ability to complete all trial procedures.

Exclusion Criteria:

1. Patients must not have had prior treatment with SHR-1210 or any other PD-L1 or PD-1 antagonists or any other oncolytic virus, and must not have had be enrolled in the phase III Study of Apatinib After Systemic Therapy in Patients With Hepatocellular Carcinoma.
2. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed.
4. Known history of hypersensitivity to any components of the SHR-1210 formulation, or M1-c6v1 (mannitol, human albumin, trehalose).
5. Active central nervous system (CNS) metastases with clinical symptoms (including cerebral edema, steroid requirement, or progressive disease). Subjects with brain or meningeal metastases that were previously treated must be clinically stable (magnetic resonance imaging [MRI] at least 4 weeks apart do not show evidence of new or enlarging metastases) and have discontinued immunosuppressive doses of systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration.
6. Patients with other malignant tumor (except cured skin basal cell carcinoma and cervical carcinoma).
7. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention, left ventricular ejection fraction(LVEF) < 50%.
8. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
9. Coagulation abnormalities (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
10. Prior systemic chemotherapy, radiotherapy, immunotherapy, hormone therapy, surgery or target therapy within 4 weeks (Or 5 half-life of the drug, calculate the longer ) before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 (with the exception of any stable chronic toxicities not expected to resolve).
11. Patients with clinical symptoms of ascites or pleural effusion, need therapeutic puncture and drainage.
12. Previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency, such as: esophageal varices, local active ulcerative lesions, gastric ulcer and duodenal ulcer, the ulcerous colitis, gastrointestinal diseases such as portal hypertension or resection of tumor with bleeding risk, etc.
13. Patients with or previous with serious hemorrhage (bleeding > 30 ml within 3 months), haemoptysis (> 5 ml within 4 weeks) of thromboembolic events within 12 months (including stroke events and/or transient ischemic attack).
14. Active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled).
15. Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, pulmonary function damaged seriously etc.
16. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or active hepatitis (transaminase does not meet the inclusion, hepatitis B virus (HBV) DNA ≥10⁴ /ml or hepatitis C virus (HCV) RNA≥103 /ml or higher); Chronic hepatitis B virus carriers who HBV DNA<2000 IU/ml(<104/ml), must receive anti-viral treatment throughout the study.
17. Participated in other clinical trials, or finish other clinical trials within 4 weeks.
18. Patients who may receive other anti-tumor systemic chemotherapy during the study.
19. Patients who has bone metastasis, have received Palliative radiotherapy (radiotherapy area > 5% marrow area).
20. Patients who may receive vaccination during the study, or previous had vaccination within 4 weeks.
21. Mental disorders history, or psychotropic drug abuse history.
22. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | From the first assignment of informed consent form up to 90 days after the last dose
  Safety as measured by the rate of TRAEs according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Overall response rate | through study completion, an average of 1 year.
Disease control rate | through study completion, an average of 1 year.
Overall survival | Up to approximately 12 months after treatment
  6 month and 12 month OS rates
Progression free survival | Up to approximately 9 months after treatment
  6 month and 9 month PFS rates

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University